CLINICAL TRIAL: NCT00786357
Title: Sleep Enhancement Training Study for Experienced Shiftworkers
Acronym: SETS-exp
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Christopher Alsten, PhD, Executive Vice President, Inner Health, Inc
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SETS-exp
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Shift-Work Sleep Disorder
Keywords: shift-work; sleep; nurse; relaxation
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: NIOSH shiftwork booklet; Behavioral: Sleep Enhancement Training System

INTERVENTIONS:
Behavioral: NIOSH shiftwork booklet — weekly readings about coping with shiftwork
Behavioral: Sleep Enhancement Training System — 4 week program of readings and relaxation programs

SUMMARY:
The purpose of this study is to determine if a modified version of the Sleep Enhancement Fatigue Reduction Training (SEFRT) system can improve sleep and health-related symptoms and quality of life in experienced shift-working nurses.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking nurses
* scheduled to work at least 2 consecutive night shifts per week during the next 3 months
* ≥40 years of age
* experiencing disturbed sleep related to night-shift

Exclusion Criteria:

* current diagnosis of sleep disorder or affective illness

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
actigraphy measures of sleep | 3 months

SECONDARY OUTCOMES:
subjective measures of sleep and well-being | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R. Alsten, PhD, Principal Investigator — Inner Health, Inc.
Locations (1):
- University of California, San Francisco, San Francisco, California, United States